CLINICAL TRIAL: NCT05290662
Title: A Prospective Multicenter Observational Study to Assess Long-term Outcome of Participants Who Have Received oNKord®
Brief Title: Registry of Patients Having Received oNKord®
Status: Recruiting | Type: Observational
Sponsor: Glycostem Therapeutics BV (Industry)
Responsible Party: Sponsor
Other Study IDs: ReKORD
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-06

CONDITIONS: AML
Keywords: NK cells; Umbilical cord blood; oNKord; Registry; Off the shelf
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants having received oNKord® as part of the WiNK clinical trial: WiNK is a Phase I/IIa trial to evaluate the safety and efficacy of oNKord® in adults with acute myeloid leukemia (AML) who are in morphologic complete remission with residual measurable disease and not currently proceeding to hematopoietic stem cell transplantation
  Interventions: Drug: oNKord®; Drug: Cyclophosphamide/Fludarabine (Cy/Flu)

INTERVENTIONS:
Drug: oNKord® — Allogeneic ex vivo-generated Natural Killer (NK) cells from CD34+ umbilical cord blood progenitor cells
Drug: Cyclophosphamide/Fludarabine (Cy/Flu) — Lymphodepleting conditioning regimen

SUMMARY:
ReKORD is an observational study (Registry) enrolling participants who have received at least one dose of oNKord® (allogeneic ex vivo-generated Natural Killer [NK] cells from CD34+ umbilical cord blood progenitor cells) in a clinical trial. Participants from multiple previous clinical trials of oNKord® can be enrolled in this Registry.

DETAILED DESCRIPTION:
To be eligible for this Registry, participants must have received at least one dose of oNKord® in a clinical trial. Eligible participants will be enrolled after signing the informed consent form (ICF). Participant characteristics, treatment history, and clinical trial outcome data at clinical trial discontinuation/completion will be collected. On a yearly basis after the last clinical trial visit, the investigator will collect the participants' medical status and enter them in the Registry database. Major clinical events, including concomitant medication or therapy, that occurred since the previous assessment will be recorded. No protocol-specific visits or interventions will be required. Participants will be followed up until 3 years after the first oNKord® infusion.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of at least one dose of oNKord® in a clinical trial
* Participation must be within 3 years after the first infusion of oNKord®
* Signature of ICF

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who have received at least one dose of oNKord® in a clinical trial and are within 3 years of follow-up after the first infusion, and who have provided informed consent for participation in this Registry.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of SAEs related to oNKord® over time | 3 years
  Safety
Incidence of SAEs related to Cyclophosphamide-Fludarabine over time | 3 years
  Safety
Long-term follow-up on survival | 3 years
Long-term follow-up on disease status | 3 years
Long-term follow-up on cancer-related treatments | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Medizinische Hochschule Hannover, Hanover, Germany
- University Hospital Basel, Basel, Switzerland